CLINICAL TRIAL: NCT03285386
Title: The Effects of Prior Exercise on Pulmonary Oxygen Uptake Kinetics and the Power-Duration Relationship in Type 1 Diabetes
Brief Title: Priming Exercise in Type 1 Diabetes
Acronym: PET1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Hope University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LiverpoolHopeUni
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants will serve as their own controls. Participants will alternate between "primed" (experimental condition) and "non-primed" (control condition) in their visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Priming Exercise (Experimental): Participants will perform constant power output tests at four separate, fixed intensities to exhaustion on a cycle ergometer on separate days. These exhaustive, constant power tests will be preceded by 3 minutes of light cycling, 6 minutes of high intensity cycling, 7 minutes of rest and 3 minutes of light cycling.
  Interventions: Behavioral: Priming exercise
- Control (Active Comparator): Participants will perform constant power output tests at four separate, fixed intensities to exhaustion on a cycle ergometer on separate days. These exhaustive, constant power tests will be preceded by 3 minutes of light cycling only.
  Interventions: Behavioral: Control Exercise

INTERVENTIONS:
Behavioral: Priming exercise — All participants will perform a bout of high-intensity "priming" exercise for 6 minutes, 10 minutes prior to undertaking an exhaustive exercise test on four separate occasions.
  Arms: Priming Exercise
Behavioral: Control Exercise — All participants will perform 3 minutes of baseline cycling prior to undertaking an exhaustive exercise test on four separate occasions.
  Arms: Control

SUMMARY:
Critical power is an important threshold in exercise physiology, and is an important determinant of the ability to tolerate high-intensity exercise. The ability to tolerate such exercise is drastically impaired in certain chronic conditions, such as type 1 diabetes. Whilst the most important physiological factors that determine critical power have yet to be determined, previous work from our laboratory suggests that it is related to the speed of oxygen uptake at the onset of exercise. This study will look to utilise "priming" exercise as an intervention to improve the speed of these oxygen uptake "kinetics", and thus critical power and exercise tolerance in individuals with type 1 diabetes. We hypothesize that oxygen uptake kinetics will be faster and critical power will be higher when exercise is performed with compared to without a prior bout of high-intensity priming exercise in a population of individuals with type 1 diabetes.

DETAILED DESCRIPTION:
The ability to tolerate high-intensity exercise, or exercise tolerance, is a key factor that can influence clinical outcomes in a range of conditions. The "critical power" is an important physiological threshold that demarcates exercise intensities that can be sustained for prolonged periods (i.e. below critical power) from intensities that result in exhaustion in a relatively short period of time (i.e. 2-30 minutes, above critical power). Critical power is therefore a key determinant of exercise tolerance. The speed with which oxygen uptake rises at the onset of exercise (i.e. oxygen uptake "kinetics") has been shown by work from our laboratory to be a key determinant of critical power. One intervention that can acutely improve the oxygen uptake kinetics is the performance of a prior bout of high-intensity exercise, known as "priming exercise". Patients with type 1 diabetes have previously been shown to have impaired exercise tolerance compared to healthy controls. The performance of priming exercise therefore represents a potential intervention to acutely improve oxygen uptake kinetics, and therefore critical power and exercise tolerance, in type 1 diabetic individuals. The purpose of this study is therefore to assess the influence of priming exercise on oxygen uptake kinetics and critical power in a population of type 1 diabetic individuals.

ELIGIBILITY:
Inclusion Criteria:

Suffering from Type 1 diabetes with a diagnosed disease duration of 2 - 20 years and no comorbidities.

Exclusion Criteria:

History of stroke, congestive heart failure, hypertension, or cardiopulmonary disease.

Current smoking or have been smoking within the last 12 months Symptomatic autonomic or distal neuropathy HbA1c > 64 mmol/mol Hypoglycaemia unawareness in the last 6 months Taking any medications other than insulin.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Critical power | 3-9 weeks
  The power asymptote of the hyperbolic relationship between power and the tolerable duration of exercise.
Phase II time constant of pulmonary oxygen uptake kinetics | 3-9 weeks
  Time taken for oxygen uptake to attain 63% of its asymptotic amplitude.
Time constant for muscle deoxygenation kinetics (assessed by near-infrared spectroscopy) | 3-9 weeks
  Time taken for muscle deoxyhaemoglobin to attain 63% of its asymptotic amplitude.

SECONDARY OUTCOMES:
W' | 3-9 weeks
  Curvature constant of the power-duration relationship. Finite work capacity available above critical power.
Time constant for heart rate kinetics | 3-9 weeks
  Time taken for heart rate to attain 63% of its asymptotic amplitude.

CONTACTS AND LOCATIONS:
Overall Officials: Richie P Goulding, Principal Investigator — Liverpool Hope University
Locations (1):
- Liverpool Hope University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymized participant data will be made available to the public in the form of research presentations and a journal article. Anonymized individual participant data not featured in either the journal article or presentations will only be made available upon request to the authors.

REFERENCES:
- [Background] Goulding RP, Roche DM, Marwood S. Prior exercise speeds pulmonary oxygen uptake kinetics and increases critical power during supine but not upright cycling. Exp Physiol. 2017 Sep 1;102(9):1158-1176. doi: 10.1113/EP086304. Epub 2017 Jul 26. PMID 28627041
- [Background] Behnke BJ, Kindig CA, McDonough P, Poole DC, Sexton WL. Dynamics of microvascular oxygen pressure during rest-contraction transition in skeletal muscle of diabetic rats. Am J Physiol Heart Circ Physiol. 2002 Sep;283(3):H926-32. doi: 10.1152/ajpheart.00059.2002. PMID 12181120
- [Background] Sexton WL, Poole DC, Mathieu-Costello O. Microcirculatory structure-function relationships in skeletal muscle of diabetic rats. Am J Physiol. 1994 Apr;266(4 Pt 2):H1502-11. doi: 10.1152/ajpheart.1994.266.4.H1502. PMID 8184927
- [Background] Kindig CA, Sexton WL, Fedde MR, Poole DC. Skeletal muscle microcirculatory structure and hemodynamics in diabetes. Respir Physiol. 1998 Feb;111(2):163-75. doi: 10.1016/s0034-5687(97)00122-9. PMID 9574868
- [Background] Burnley M, Davison G, Baker JR. Effects of priming exercise on VO2 kinetics and the power-duration relationship. Med Sci Sports Exerc. 2011 Nov;43(11):2171-9. doi: 10.1249/MSS.0b013e31821ff26d. PMID 21552161